CLINICAL TRIAL: NCT00618241
Title: The Influence of Raltegravir (MK-0518) on the Pharmacokinetics of Single-dose Lamotrigine in Healthy Male Subjects (GRANOLA)
Brief Title: Pharmacokinetic Study on Raltegravir and Lamotrigine
Acronym: GRANOLA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr. D.M. Burger, hospital pharmacist, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 07.06
Record Dates: First submitted 2008-02-05; First posted 2008-02-19 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2011-05

CONDITIONS: HIV Infection
Keywords: interactions; neuropathic pain; pharmacokinetics
MeSH Terms: conditions — HIV Infections; Neuralgia | interventions — Lamotrigine; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Group A: day 1-5 Raltegravir 400 mg oral BD (twice daily). Lamotrigine one oral dose 100 mg on day 4. Wash-out 6-31. Followed by one oral dose Lamotrigine 100 mg on day 34.
  5 days Raltegravir 400 mg oral BD. Lamotrigine one oral dose 100mg on day 34.
  Interventions: Drug: lamotrigine; Drug: Raltegravir
- B (Active Comparator): Group B: day 4 Lamotrigine one oral dose on day 4. Wash-out day 6-28 followed by Raltegravir 400 mg oral BD day 29-33. One dose Lamotrigine 100 mg oral on day 32.
  One dose Lamotrigine 100 mg oral.
  Interventions: Drug: lamotrigine; Drug: Raltegravir

INTERVENTIONS:
Drug: lamotrigine — 100 mg
  Other Names: Lamictal
Drug: Raltegravir — 400 mg BD

SUMMARY:
The purpose of this study is to determine whether interactions between raltegravir and lamotrigine take place and to study the safety of the combination raltegravir/lamotrigine before used in HIV patients.

DETAILED DESCRIPTION:
Lamotrigine is an anticonvulsive drug that is used both for the treatment of HIV-associated neuropathic pain and the treatment of epilepsy in HIV-infected individuals. Lamotrigine is metabolized via glucuronidation.

Raltegravir is a newly developed integrase inhibitor that is also metabolized via glucuronidation.

Since both agents are metabolized via glucuronidation, there is a possibility of competition for glucuronidation, leading to drug-drug interactions between raltegravir and lamotrigine.

This primary objective of this study is to determine the effect of raltegravir on the pharmacokinetics of single dose lamotrigine (by intrasubject comparison). A secondary objective is to determine the effect of single dose lamotrigine on the pharmacokinetics of raltegravir when compared to historical controls. Another secondary objective is to evaluate the safety of combined use of single dose lamotrigine and raltegravir.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age
* Subject does not smoke more than 10 cigarettes, 2 cigars or 2 pipes per day
* Subject has a Quetelet Index of 18 to 30 kg/m2
* Subject is able and willing to sign informed consent
* Subject is in good age-appropriate health condition
* Subject has a normal blood pressure and pulse rate

Exclusion Criteria:

* History of sensitivity/idiosyncrasy to medicinal products or excipients
* Positive HIV test
* Positive hepatitis B or C test
* Therapy with any drug (2 weeks preceding dosing) except for paracetamol
* Relevant history or presence of pulmonary disorders, cardiovascular
* History of or current abuse of drugs, alcohol or solvents
* Inability to understand the nature and extent of the trial and procedures
* Participation in a drug trial within 60 days prior to the first dose
* Donation of blood within 60 days prior to the first dose
* Febrile illness within 3 days before the first dose

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of lamotrigine, lamotrigine-2N-glucuronide, and raltregravir | just before dosing, at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 24 hours and 48 hours after dosing on study days 4-5 and 32-33.

SECONDARY OUTCOMES:
Determination of pharmacokinetic parameters (AUC, Cmax, Tmax, Cmin and T 1/2) by noncompartmental analysis | at each sampling time

CONTACTS AND LOCATIONS:
Overall Officials: David M. Burger, PharmD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] van Luin M, Colbers A, Verwey-van Wissen CP, van Ewijk-Beneken-Kolmer EW, van der Kolk M, Hoitsma A, da Silva HG, Burger DM. The effect of raltegravir on the glucuronidation of lamotrigine. J Clin Pharmacol. 2009 Oct;49(10):1220-7. doi: 10.1177/0091270009345689. Epub 2009 Aug 28. PMID 19717722
- See also: Results published in The Journal of Clinical Pharmacology; 2009; 49; 1220 — https://pubmed.ncbi.nlm.nih.gov/19717722/